CLINICAL TRIAL: NCT04081467
Title: MARS-PRE: MARcatori Biologici e Funzionali Per la Biomedicina aStronautica di PREcisione
Brief Title: Biological and Functional Markers for Precision Astronautical Biomedicine
Acronym: MARS-PRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science and Research Centre Koper (Other)
Collaborators: University of Padova (Other); University of Bari (Other); University of Genova (Other); University of L'Aquila (Other); University of Pavia (Other); University of Trieste (Other); Humanitas Hospital, Italy (Other); University of Rome (Unknown)
Responsible Party: Principal Investigator, Rado Pisot, prof. Rado Pisot, PhD, prof. Marco Narici, MD, PhD, prof. Bostjan Simunic, PhD, Assistant professor Uros Marusic, PhD,, Science and Research Centre Koper
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR2019 MARS-PRE
Record Dates: First submitted 2019-07-31; First posted 2019-09-09 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy | interventions — Bed Rest; Immobilization

STUDY DESIGN:
Intervention Model Description: One group of 10 will undergo 10 days of horizontal bed rest without countermeasures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bed rest condition (Experimental): Bed rest condition without any additional intervention
  Interventions: Other: Bed rest

INTERVENTIONS:
Other: Bed rest — 10-day of complete bed rest
  Other Names: immobilization; bed rest confinement; prolonged physical inactivity

SUMMARY:
In the current study the investigators will study early biomarkers of human degradation. In 10-day horizontal bed rest the investigators will enroll 10 healthy male subjects (18-30years, BMI 20-28kg/m2). Pre-, mid- and post-bed rest the investigators will perform various measurements, some of them will be invasive (blood samples and muscle biopsies), which will be carefully taken by the medical staff. The subjects will be placed in hospital rooms and have 24-hour medical supervision, adequate hygiene, nutrition, passive exercise, entertainment and visits.

DETAILED DESCRIPTION:
Ten young male participants will undergo 10 days of horizontal bed rest. Before, during and after the investigators will monitor many biomechanical, metabolic, cardiovascular, biochemical responses.

During the bed rest period there will be no interventions. subjects will be allowed to rotate freely, with no vertical stimulus of any-kind.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 20 - 28 kg/m2
* male participants
* a healthy individual who is able to complete all the tests planned in the research protocol

Exclusion Criteria:

* smoking;
* regular alcohol consumption;
* ferromagnetic implants;
* history of deep vein thrombosis with D-dimer > 500 μg·L-1;
* acute or chronic skeletal, neuromuscular, psychological, metabolic and cardiovascular disease conditions.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Change in mittochondria respiration rate | At baseline and after 10-day bed rest
  Change in Mittochondria oxygen respiration rate per mg of muscle tissue after 10-day bed rest
Change in skeletal muscle single fibre force (in micro Newtons) | At baseline and after 10-day bed rest
  In each aprticipants at each time point approx 10 intact muscle fibres will be studied for their force production after 10-day bed rest. Isometric muscle fibre force (in mNewton) will be measured isometric force (Fo) in four subsequent maximal activations (pCa, 4.6; sarcomere length, 2.6 micrometers; temperature 12 degrees C) using an electrical motor with force transducer mounted on it.
Change in Neurological outcomes - nerve conduction velocity | At baseline and after 10-day bed rest
  Change in nerve conduction velocity after 10-day bed rest
Change in Neurological outcomes - fMRI | At baseline and after 10-day bed rest
  Change in ability to mentally imagine/perform locomotory tasks (voxel-based network analyses) after 10-day bed rest
Change in Neurological outcomes - neurocognitive assessment | At baseline and after 10-day bed rest
  Change in EEG and neurocognitive tasks parameters (event related potential; P300 component during Stroop task) after 10-day bed rest
Change in skeletal muscle NCAM expression in single fibres | Before, at day 5 and day 10 of bed rest
  Neural cell adhesion molecule (NCAM) expression will be analysed in vastus lateralis biopsy samples at three time points.

SECONDARY OUTCOMES:
Change in muscle volume after 10-day bed rest | At baseline and after 10-day bed rest
  Thigh muscle volume will be assessed by continous section obtained by 3T MRI. Muscle segmentation will done by Matlab routine.
Change in peak aerobic power after 10-day bed rest | At baseline and after 10-day bed rest
  Change in peak aerobic power (maximal oxygen consumption) will be assessed on a cycloergometer using graded load protocol.
Nonhomogeneous change in skeletal muscle pennation angle after 10-day bed rest | At baseline, every 2 days of bed rest and after 10-day bed rest
  Change in Muscle architecture will be assessed in vastus lateralis, biceps femoris, tibialis anterior, multifidus using sonography. Specifically, we will assess all three architecture parameters (pennation angle, fascicle length and thickness), however for the purspose of this outcome we hypothesize non-homogenous change throughout the whole muscles in pennation angle. The assessment will be performed before, every 2 days of bed rest and post bed rest.
Change in maximal displacement after twitch contraction after 10-day bed rest | At baseline, every 2 days of bed rest and after 10-day bed rest
  Using tensiomyography we will assess contraction time and maximal discplacement in vastus lateralis, tibialis anterior, biceps femoris, multifidus muscles. We expect that contraction time will remained the same but maximal diasplacement - a measure of a muscle tone, will increase much before the changes in muscle thickness - assessed by sonography. The assessment will be performed before, every 2 days of bed rest and post bed rest.
Change in skeletal composition after 10-day bed rest | At baseline, day 5 and after 10-day bed rest
  Using electrophoresis we will assess changes in myosing heavy chains somposition in the biopsies obtained from vastus lateralis muscle before, at day 5 and post 10 days of bed rest
Change in skeletal muscle maximal voluntary contraction after 10-day bed rest | At baseline and after 10-day bed rest
  Maximal voluntary isometric knee extensors contraction will be measured using dnamometer set at 90 deg flexion.
Change in balance after 10-day bed rest | At baseline and after 10-day bed rest
  Change in static and dynamic balance will be assessed by functional tests (gait assessed with Optogait system and balance assessed with Tensiometric plate-COP) after 10-day bed rest
Change in orthostatic tolerance after 10-day bed rest | At baseline and after 10-day bed rest
  Change in mean arterial pressure during supine-to-stand test (mmHg) will be assessed by supine to stand test, where subjects will stay 10 minutes in each position.

CONTACTS AND LOCATIONS:
Locations (1):
- Splosna bolnisnica Izola (Hospital of Izola), Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No
The data is shared among partners for various publications

REFERENCES:
- [Background] Pisot R, Marusic U, Biolo G, Mazzucco S, Lazzer S, Grassi B, Reggiani C, Toniolo L, di Prampero PE, Passaro A, Narici M, Mohammed S, Rittweger J, Gasparini M, Gabrijelcic Blenkus M, Simunic B. Greater loss in muscle mass and function but smaller metabolic alterations in older compared with younger men following 2 wk of bed rest and recovery. J Appl Physiol (1985). 2016 Apr 15;120(8):922-9. doi: 10.1152/japplphysiol.00858.2015. Epub 2016 Jan 28. PMID 26823343
- [Background] Simunic B, Koren K, Rittweger J, Lazzer S, Reggiani C, Rejc E, Pisot R, Narici M, Degens H. Tensiomyography detects early hallmarks of bed-rest-induced atrophy before changes in muscle architecture. J Appl Physiol (1985). 2019 Apr 1;126(4):815-822. doi: 10.1152/japplphysiol.00880.2018. Epub 2019 Jan 24. PMID 30676871
- [Background] Floreani M, Rejc E, Taboga P, Ganzini A, Pisot R, Simunic B, Biolo G, Reggiani C, Passaro A, Narici M, Rittweger J, di Prampero PE, Lazzer S. Effects of 14 days of bed rest and following physical training on metabolic cost, mechanical work, and efficiency during walking in older and young healthy males. PLoS One. 2018 Mar 12;13(3):e0194291. doi: 10.1371/journal.pone.0194291. eCollection 2018. PMID 29529070
- [Background] Rejc E, Floreani M, Taboga P, Botter A, Toniolo L, Cancellara L, Narici M, Simunic B, Pisot R, Biolo G, Passaro A, Rittweger J, Reggiani C, Lazzer S. Loss of maximal explosive power of lower limbs after 2 weeks of disuse and incomplete recovery after retraining in older adults. J Physiol. 2018 Feb 15;596(4):647-665. doi: 10.1113/JP274772. Epub 2018 Jan 19. PMID 29266264
- [Background] Passaro A, Soavi C, Marusic U, Rejc E, Sanz JM, Morieri ML, Nora ED, Kavcic V, Narici MV, Reggiani C, Biolo G, Zuliani G, Lazzer S, Pisot R. Computerized cognitive training and brain derived neurotrophic factor during bed rest: mechanisms to protect individual during acute stress. Aging (Albany NY). 2017 Feb 3;9(2):393-407. doi: 10.18632/aging.101166. PMID 28161695
- [Background] Marusic U, Giordani B, Moffat SD, Petric M, Dolenc P, Pisot R, Kavcic V. Computerized cognitive training during physical inactivity improves executive functioning in older adults. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2018 Jan;25(1):49-69. doi: 10.1080/13825585.2016.1263724. Epub 2016 Dec 12. PMID 27937138
- [Background] Marusic U, Kavcic V, Giordani B, Gerzevic M, Meeusen R, Pisot R. Computerized spatial navigation training during 14 days of bed rest in healthy older adult men: Effect on gait performance. Psychol Aging. 2015 Jun;30(2):334-340. doi: 10.1037/pag0000021. Epub 2015 May 4. PMID 25938245
- [Background] Marusic U, Meeusen R, Pisot R, Kavcic V. The brain in micro- and hypergravity: the effects of changing gravity on the brain electrocortical activity. Eur J Sport Sci. 2014;14(8):813-22. doi: 10.1080/17461391.2014.908959. Epub 2014 Apr 15. PMID 24734884
- [Background] Rejc E, di Prampero PE, Lazzer S, Grassi B, Simunic B, Pisot R, Antonutto G, Narici M. A 35-day bed rest does not alter the bilateral deficit of the lower limbs during explosive efforts. Eur J Appl Physiol. 2015 Jun;115(6):1323-30. doi: 10.1007/s00421-015-3111-2. Epub 2015 Jan 23. PMID 25613402